CLINICAL TRIAL: NCT03815240
Title: Comparing the Effects of Three Different Dressings on the Cutaneous Response to Pressure and Shear of Sacral Skin: an Exploratory Crossover Study
Brief Title: Comparing the Effects of Three Different Dressings on the Cutaneous Response of Sacral Skin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, PD Dr. Jan Kottner, Principal Investigator, Charite University, Berlin, Germany
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: CRC-SP-A-32
Record Dates: First submitted 2019-01-16; First posted 2019-01-24 (Actual); Results first posted 2020-05-06 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-04

CONDITIONS: Pressure Ulcer Prevention
Keywords: Pressure Ulcer Prevention; Preventive Dressings

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- no dressing (A) (Other): No dressing will be applied at sacrum before 3.5 hours loading period in supine position
  Interventions: Other: No dressing
- Mepilex (B) (Active Comparator): 'Mepilex® Border Sacrum' dressing will be applied at sacrum before 3.5 hours loading period in supine position
  Interventions: Other: Mepilex® Border Sacrum
- Allevyn (C) (Active Comparator): 'ALLEVYN Life Sacrum' dressing will be applied at sacrum before 3.5 hours loading period in supine position
  Interventions: Other: ALLEVYN Life Sacrum
- Optifaom (D) (Active Comparator): 'Optifoam® Gentle Sacrum' Dressing will be applied at sacrum before 3.5 hours loading period in supine position
  Interventions: Other: Optifoam® Gentle Sacrum

INTERVENTIONS:
Other: No dressing — no dressing at sacrum
  Arms: no dressing (A)
Other: Mepilex® Border Sacrum — adhesive sacrum dressing
  Arms: Mepilex (B)
Other: ALLEVYN Life Sacrum — adhesive sacrum dressing
  Arms: Allevyn (C)
Other: Optifoam® Gentle Sacrum — adhesive sacrum dressing
  Arms: Optifaom (D)

SUMMARY:
Skin functional parameters such as erythema or stratum corneum hydration have been successfully used in PU prevention research. These parameters are able to discriminate effects of different loading intensities and to measure PU preventive device performance.

The overall aim of this study is to measure the effects of Mepilex® Border Sacrum Dressing on the skin structure and function during mechanical loading compared to (1) no dressing, (2) ALLEVYN Life Sacrum Dressing and (3) Optifoam® Gentle Liquitrap Sacrum Dressing.

DETAILED DESCRIPTION:
Pressure ulcers (PUs) are severe and unwanted cutaneous lesions and subcutaneous wounds caused by prolonged skin and underlying soft tissue deformation. In the supine position they predominantly occur near to bony prominences, like at the sacral area. The cornerstone of PU prevention is repositioning, early mobilization and the use of special support surfaces. In addition, empirical evidence suggests that the application of preventive dressings on PU predilection sites helps to prevent PU development.

Skin functional parameters such as erythema or stratum corneum hydration have been successfully used in PU prevention research. These parameters are able to discriminate effects of different loading intensities and to measure PU preventive device performance. Recently it could be shown that there are associations between structural and functional skin changes at the sacral area during loading. The overall aim of this study is to measure the effects of Mepilex® Border Sacrum Dressing on the skin structure and function during mechanical loading compared to no dressing, ALLEVYN Life Sacrum and Optifoam® Gentle Liquitrap Sacrum.

The procedure of one visit will be as follows:

After a skin acclimatization time of 30 minutes baseline measurements and Cyanoacrylate Skin Surface (CSSS)-stripping will be performed. Then a randomization envelope will be opened and the corresponding dressing will be applied or the skin will be left uncovered. The subject will then lie in supine position on a standard hospital mattress for a loading period of 3.5 hours. Every 30 minutes the head of the bed will be elevated to 45° for five minutes. During these five minutes, the participants will be instructed to bend their knees and to drag the feet repeatedly forth and back 10 times in order to simulate shear forces. The whole exercise will be done six times, after 0.5, 1, 1.5, 2, 2.5 and 3 hours. After 3.5 hours loading time in supine position the subjects will move into prone position. The dressing (if present) will be removed and all skin measurements and CSSS-stripping will be conducted again. The subjects will come back for another three times completing the remaining interventions. At the end, each volunteer will have received all three types of dressings once and once no dressing. In between, there are at least 3 weeks to prevent possible carry over effects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female volunteers
* 65 to 80 years
* Body Mass Index 18.5 to 29.9 kg/m2
* Non-smoker of at least one year (including electronic-cigarettes)
* Informed consent
* Being free of any clinical dermatosis in the investigational area
* Intact sacral skin without scars
* Skin phototype I, II, or III (according to Fitzpatrick)
* No regular use of leave-on products on the sacral skin
* Willing and able to fulfil the study requirements

Exclusion Criteria:

* Disability to maintain in supine or prone Position
* Acute diseases
* Known hyper-sensibility or allergy to the study product or any of its ingredients
* Extensive UV exposure 4 weeks before study inclusion
* Use of topical treatment on the investigational areas or systemic Treatment within the 4 past weeks (topical hyaluronan, anti-inflammatory drugs, corticoids, retinoids, NSIDS etc.) that would interfere with assessment and/or investigational treatments
* Medical history of skin cancer
* History of established Diabetes mellitus, cardiac or renal insufficiency, COPD
* Chronic inflammatory skin disorders such as atopic dermatitis, psoriasis, lichen planus
* Participation in another study 4 weeks prior to study start

Ages: 65 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-02-08 (Actual); Primary Completion 2019-07-23 (Actual); Study Completion 2019-07-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Charité-Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study took place at the Clinical Research Center for Hair and Skin Science in Berlin, Germany from January 2019 to July 2019 and involved 12 healthy female volunteers
Groups:
- No Dressing, Mepilex, Allevyn, Optifoam: Dressing application order:
  no dressing (A), Mepilex® Border Sacrum (B), ALLEVYN Life Sacrum (C), Optifoam® Gentle Sacrum (D)
- Mepilex, no Dressing, Optifoam, Allevyn: Dressing application order:
  Mepilex® Border Sacrum (B), no dressing (A), Optifoam® Gentle Sacrum (D), ALLEVYN Life Sacrum (C)
- No Dressing, Mepilex, Optifoam, Allevyn: Dressing application order:
  no dressing (A), Mepilex® Border Sacrum (B), Optifoam® Gentle Sacrum (D), ALLEVYN Life Sacrum (C)
- No Dressing, Allevyn, Mepilex, Optifoam: Dressing application order:
  no dressing (A), ALLEVYN Life Sacrum (C), Mepilex® Border Sacrum (B), Optifoam® Gentle Sacrum (D)
- Optifoam, Allevyn, no Dressing, Mepilex: Dressing application order:
  Optifoam® Gentle Sacrum (D), ALLEVYN Life Sacrum (C), no dressing (A), Mepilex® Border Sacrum (B)
- Optifoam, Mepilex, Allevyn, no Dressing,: Dressing application order:
  Optifoam® Gentle Sacrum (D), Mepilex® Border Sacrum (B), ALLEVYN Life Sacrum (C), no dressing (A)
- Mepilex, Optifoam, no Dressing, Allevyn: Dressing application order:
  Mepilex® Border Sacrum (B), Optifoam® Gentle Sacrum (D), no dressing (A), ALLEVYN Life Sacrum (C)
- Allevyn, no Dressing, Mepilex, Optifoam: Dressing application order:
  ALLEVYN Life Sacrum (C), no dressing (A), Mepilex® Border Sacrum (B), Optifoam® Gentle Sacrum (D)
- Optifoam, Allevyn, Mepilex, no Dressing: Dressing application order:
  Optifoam® Gentle Sacrum (D), ALLEVYN Life Sacrum (C), Mepilex® Border Sacrum (B), no dressing (A)
Period: Intervention no Dressing
Arm/Group | No Dressing, Mepilex, Allevyn, Optifoam | Mepilex, no Dressing, Optifoam, Allevyn | No Dressing, Mepilex, Optifoam, Allevyn | No Dressing, Allevyn, Mepilex, Optifoam | Optifoam, Allevyn, no Dressing, Mepilex | Optifoam, Mepilex, Allevyn, no Dressing, | Mepilex, Optifoam, no Dressing, Allevyn | Allevyn, no Dressing, Mepilex, Optifoam | Optifoam, Allevyn, Mepilex, no Dressing
Started (Cross-over study. Each of the 12 participants received each intervention once (total number is 12).) | 2 | 1 | 1 | 2 | 1 | 2 | 1 | 1 | 1
Completed (Cross-over study. Each of the 12 participants received each intervention once (total number is 12).) | 2 | 1 | 1 | 2 | 1 | 2 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Intervention Mepilex Dressing
Arm/Group | No Dressing, Mepilex, Allevyn, Optifoam | Mepilex, no Dressing, Optifoam, Allevyn | No Dressing, Mepilex, Optifoam, Allevyn | No Dressing, Allevyn, Mepilex, Optifoam | Optifoam, Allevyn, no Dressing, Mepilex | Optifoam, Mepilex, Allevyn, no Dressing, | Mepilex, Optifoam, no Dressing, Allevyn | Allevyn, no Dressing, Mepilex, Optifoam | Optifoam, Allevyn, Mepilex, no Dressing
Started (Cross-over study. Each of the 12 participants received each intervention once (total number is 12).) | 2 | 1 | 1 | 2 | 1 | 2 | 1 | 1 | 1
Completed (Cross-over study. Each of the 12 participants received each intervention once (total number is 12).) | 2 | 1 | 1 | 2 | 1 | 2 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Intervention Allevyn Dressing
Arm/Group | No Dressing, Mepilex, Allevyn, Optifoam | Mepilex, no Dressing, Optifoam, Allevyn | No Dressing, Mepilex, Optifoam, Allevyn | No Dressing, Allevyn, Mepilex, Optifoam | Optifoam, Allevyn, no Dressing, Mepilex | Optifoam, Mepilex, Allevyn, no Dressing, | Mepilex, Optifoam, no Dressing, Allevyn | Allevyn, no Dressing, Mepilex, Optifoam | Optifoam, Allevyn, Mepilex, no Dressing
Started (Cross-over study. Each of the 12 participants received each intervention once (total number is 12).) | 2 | 1 | 1 | 2 | 1 | 2 | 1 | 1 | 1
Completed (Cross-over study. Each of the 12 participants received each intervention once (total number is 12).) | 2 | 1 | 1 | 2 | 1 | 2 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Intervention Optifoam Dressing
Arm/Group | No Dressing, Mepilex, Allevyn, Optifoam | Mepilex, no Dressing, Optifoam, Allevyn | No Dressing, Mepilex, Optifoam, Allevyn | No Dressing, Allevyn, Mepilex, Optifoam | Optifoam, Allevyn, no Dressing, Mepilex | Optifoam, Mepilex, Allevyn, no Dressing, | Mepilex, Optifoam, no Dressing, Allevyn | Allevyn, no Dressing, Mepilex, Optifoam | Optifoam, Allevyn, Mepilex, no Dressing
Started (Cross-over study. Each of the 12 participants received each intervention once (total number is 12).) | 2 | 1 | 1 | 2 | 1 | 2 | 1 | 1 | 1
Completed (Cross-over study. Each of the 12 participants received each intervention once (total number is 12).) | 2 | 1 | 1 | 2 | 1 | 2 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 12 female participants between 65 to 80 years.
Groups:
- no Dressing, Mepilex, Allevyn, Optifoam (in Different Order): Cross-over study. Each of the 12 participants received each intervention once (no dressing, Mepilex® Border Sacrum, ALLEVYN Life Sacrum, Optifoam® Gentle Sacrum)
Arm/Group | no Dressing, Mepilex, Allevyn, Optifoam (in Different Order)
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.2 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Germany | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in Skin Surface Temperature From Baseline
Description: A skin thermometer based on infrared technique (Courage and Khazaka Electronic GmbH) was used to measure the skin surface temperature at the sacrum
Time Frame: Change from baseline after 3.5 hours loading period at visit 1 (Day 0), visit 2 (not before 3 weeks after visit 1), visit 3 (not before 3 weeks after visit 2), visit 4 (not before 3 weeks after visit 3).
Population: Cross-over study. Each of the 12 participants received each intervention once (total number is 12).
Measure: Median (Inter-Quartile Range); unit: °C
Groups:
- no Dressing (A): No dressing was applied at sacrum before 3.5 hours loading period in supine position
- Mepilex (B): 'Mepilex® Border Sacrum' dressing was applied at sacrum before 3.5 hours loading period in supine position
- Allevyn (C): 'ALLEVYN Life Sacrum' dressing was applied at sacrum before 3.5 hours loading period in supine position
- Optifaom (D): 'Optifoam® Gentle Sacrum' Dressing was applied at sacrum before 3.5 hours loading period in supine position
Arm/Group | no Dressing (A) | Mepilex (B) | Allevyn (C) | Optifaom (D)
Number analyzed (Participants) | 12 | 12 | 12 | 12
°C | 3.1 [1.9 to 4.1] | 3.8 [2.8 to 4.1] | 3.0 [2.4 to 4.4] | 3.3 [2.3 to 3.9]

2. Primary Outcome: Change in Stratum Corneum Hydration (SCH) From Baseline
Description: Corneometer CM 825 (Courage and Khazaka Electronic GmbH) was used to measure the stratum corneum hydration (SCH) at the sacrum in arbitrary units (AU) (range 0-120 AU). Lower values represent reduced skin hydration in the upper skin layer. The measurement is based on capacitance measurement of a dielectric medium. The change in the dielectric constant due to skin surface hydration by capacitance differences of a precision capacitor is measured.
Time Frame: as for outcome 1
Population: Cross-over study. Each of the 12 participants received each intervention once (total number is 12).
Measure: Median (Inter-Quartile Range); unit: arbitrary units
Arm/Group | no Dressing (A) | Mepilex (B) | Allevyn (C) | Optifaom (D)
Number analyzed (Participants) | 12 | 12 | 12 | 12
arbitrary units | 7.0 [0.7 to 13.3] | 4.4 [1.2 to 11.5] | 5.9 [-0.4 to 9.2] | 7.3 [3.6 to 15.0]

3. Primary Outcome: Change in Erythema Index (EI) From Baseline
Description: Mexameter MX18 (Courage and Khazaka Electronic GmbH) was used to measure the Erythema index at the sacrum. This device uses specific wavelengths (the intensity of the reflected red (λ = 660 nm) and green (λ = 568 nm) lights) to measure the absorption capacity of the skin (specifically the content of hemoglobin in the skin) and presents values from 0 to 999. Lower values represent less redness.
Time Frame: as for outcome 1
Population: Cross-over study. Each of the 12 participants received each intervention once (total number is 12).
Measure: Median (Inter-Quartile Range); unit: arbitrary units
Arm/Group | no Dressing (A) | Mepilex (B) | Allevyn (C) | Optifaom (D)
Number analyzed (Participants) | 12 | 12 | 12 | 12
arbitrary units | 29 [19 to 49] | 7 [-9 to 45] | 41 [-2 to 63] | 4 [-24 to 25]

4. Primary Outcome: Change in Average Roughness (Rz) From Baseline
Description: The Visioscan VC 98 camera (Courage and Khazaka Electronic GmbH) was used to capture images of the sacrum. The special LED UV light source with diffuser provides sharp, very high resolution images of the skin surface (255 grey levels representing different depths). The grey level distribution allows the calculation of different roughness parameters to quantitatively describe the skin surface.
Time Frame: as for outcome 1
Population: Cross-over study. Each of the 12 participants received each intervention once (total number is 12).
Measure: Median (Inter-Quartile Range); unit: micrometre
Arm/Group | no Dressing (A) | Mepilex (B) | Allevyn (C) | Optifaom (D)
Number analyzed (Participants) | 12 | 12 | 12 | 12
micrometre | -0.8 [-7.6 to 1.8] | -1 [-5.3 to 2.8] | -0.8 [-2.0 to 0.9] | -6.3 [-9.4 to -5.0]

5. Primary Outcome: Change in Arithmetic Average Roughness (Ra) From Baseline
Description: as for outcome 4
Time Frame: as for outcome 1
Population: Cross-over study. Each of the 12 participants received each intervention once (total number is 12).
Measure: Median (Inter-Quartile Range); unit: micrometre
Arm/Group | no Dressing (A) | Mepilex (B) | Allevyn (C) | Optifaom (D)
Number analyzed (Participants) | 12 | 12 | 12 | 12
micrometre | -0.8 [-3.9 to 2.4] | -0.3 [-5.8 to 3.1] | 0.5 [-0.5 to 2.3] | -4.5 [-6.9 to -0.6]

6. Primary Outcome: Change in Maximum Roughness (Rmax) From Baseline
Description: as for outcome 4
Time Frame: as for outcome 1
Population: Cross-over study. Each of the 12 participants received each intervention once (total number is 12).
Measure: Median (Inter-Quartile Range); unit: micrometre
Arm/Group | no Dressing (A) | Mepilex (B) | Allevyn (C) | Optifaom (D)
Number analyzed (Participants) | 12 | 12 | 12 | 12
micrometre | -0.5 [-8.8 to 2.6] | -1.8 [-7.8 to 2.4] | -1.3 [-3.1 to 1.0] | -8.0 [-12.3 to -5.1]

7. Primary Outcome: Change in Interleukin IL-1alpha Concentration From Baseline
Description: Based on Cyanoacrylate Skin Surface (CSSS)-Stripping, corneocytes was collected in order to analyse changes regarding interleukin IL-1alpha concentrations.
Time Frame: as for outcome 1
Population: Cross-over study. Each of the 12 participants received each intervention once (total number is 12).
Measure: Median (Inter-Quartile Range); unit: picogramme/microgramme
Arm/Group | no Dressing (A) | Mepilex (B) | Allevyn (C) | Optifaom (D)
Number analyzed (Participants) | 12 | 12 | 12 | 12
picogramme/microgramme | 1.1 [-0.1 to 4.2] | -0.1 [-0.9 to 2.5] | 1.3 [0.1 to 3.7] | 1.3 [-0.8 to 2.8]

8. Secondary Outcome: Occurence of Sacral Pain
Description: The occurrence of pain (yes/no)
Time Frame: Captured from baseline until the end of the loading period after 3.5 hours at visit 1 (Day 0), visit 2 (not before 3 weeks after visit 1), visit 3 (not before 3 weeks after visit 2), visit 4 (not before 3 weeks after visit 3).
Population: Cross-over study. Each of the 12 participants received each intervention once (total number is 12).
Measure: Count of Participants; unit: Participants
Groups:
- Optifoam (D): 'Optifoam® Gentle Sacrum' Dressing was applied at sacrum before 3.5 hours loading period in supine position
Arm/Group | no Dressing (A) | Mepilex (B) | Allevyn (C) | Optifoam (D)
Number analyzed (Participants) | 12 | 12 | 12 | 12
Participants | 0 | 0 | 0 | 0

9. Secondary Outcome: Time Until First Reporting of Sacral Pain
Description: Time from baseline until the subject reported pain at sacrum
Time Frame: Sacral pain was assessed from baseline up until 3.5 hours loading period at visit 1 (Day 0), visit 2 (not before 3 weeks after visit 1), visit 3 (not before 3 weeks after visit 2), visit 4 (not before 3 weeks after visit 3).
Population: Cross-over study. Each of the 12 participants received each intervention once (total number is 12).
Measure: Median (Inter-Quartile Range); unit: minutes
Groups:
- Optofoam (D): 'Optifoam® Gentle Sacrum' Dressing was applied at sacrum before 3.5 hours loading period in supine position
Arm/Group | no Dressing (A) | Mepilex (B) | Allevyn (C) | Optofoam (D)
Number analyzed (Participants) | 12 | 12 | 12 | 12
minutes | NA [NA to NA] — no participant experienced pain during the study visits | NA [NA to NA] — no participant experienced pain during the study visits | NA [NA to NA] — no participant experienced pain during the study visits | NA [NA to NA] — no participant experienced pain during the study visits

10. Secondary Outcome: Change in Erythema Score From Baseline
Description: Erythema was assessed by visual inspection. A metric scale will be used: 0 = none 1 = mild (slight reddening), 2 = moderate (distinct redness), 3 = severe (strong redness, dark red)
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | no Dressing (A) | Mepilex (B) | Allevyn (C) | Optifaom (D)
Number analyzed (Participants) | 12 | 12 | 12 | 12
Participants
  no erythema | 9 | 6 | 5 | 5
  mild erythema | 3 | 6 | 6 | 5
  moderate erythema | 0 | 0 | 1 | 2

ADVERSE EVENTS:
Time Frame: during each visit (four visits per subject), 5.5 hours each
Arm/Group | no Dressing (A) | Mepilex (B) | Allevyn (C) | Optifoam (D)
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-15): https://cdn.clinicaltrials.gov/large-docs/40/NCT03815240/Prot_SAP_000.pdf